CLINICAL TRIAL: NCT06485661
Title: Intermediate Term Effect of Captopril on Left Ventricle Global Longitudinal Strain in Patients With Duchenne Myodystrophy
Brief Title: Effect of Captopril on GLS in Duchenne Myodystrophy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS180/2024
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-06

CONDITIONS: Effect of Drug
MeSH Terms: interventions — Captopril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Duchenne patients subjected to captopril (Other)
  Interventions: Drug: Captopril Tablets

INTERVENTIONS:
Drug: Captopril Tablets — Patients will be given captopril to see effect on global longitudinal strain

SUMMARY:
To outline the intermediate term effect of prescribing Captopril as an add on therapy on Left ventricular functions as measured by Global longitudinal strain in patients with Duchenne myodystrophy (DMD)

DETAILED DESCRIPTION:
ACEI slowing down the onset and the progression of dystrophinopathic cardiomyopathy.

To outline the intermediate term effect of prescribing Captopril as an add on therapy on Left ventricular functions as measured by Global longitudinal strain in patients with Duchenne myodystrophy (DMD

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed Duchenne myodystrophy (DMD) patients with abnormal GLS < -18% with minimum age of 6 years old.

Exclusion Criteria:

* Any patient who refuses to sign an informed consent.
* Contraindication to ACEI: hypersensitivity - renal impairment - bilateral renal artery stenosis - aortic valve stenosis - hyperkalemia - hypotension.
* Reduced ejection fraction below 50%.

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
The impaired global longitudinal strain will change in echo in the number of participants with duchenne myodystrophy | 6 months
  Impaired Global longitudinal strain will be changed in echo after 6 months of treatment with Captopril in patients with duchenne myodystrophy

CONTACTS AND LOCATIONS:
Overall Officials: Mona Mostafa Rayan, MD, Principal Investigator — Professor of cardiology -Ain Shams university
Locations (1):
- Ain Shams university, Cairo, Egypt